CLINICAL TRIAL: NCT06678256
Title: Pregnancy Outcomes in Patients With Adult Congenital Heart Disease
Brief Title: A Study of Pregnancy Outcomes in Congenital Heart Disease
Acronym: POACHD
Status: Suspended | Type: Observational
Why Stopped: Suspended due to delayed procurement of equipment.
Sponsor: Mayo Clinic (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Alexander C. Egbe, Principal Investigator, Mayo Clinic
Other Study IDs: 24-007434; 5R01HL160761-04 (NIH)
Record Dates: First submitted 2024-11-05; First posted 2024-11-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Congenital Heart Disease
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to determine if a biomarker assay obtained peripartum (1st-3rd trimester and post-partum) in patients with adult congenital heart disease can predict future risk of cardiovascular adverse events and determine if temporal changes in biomarkers levels throughout the peripartum period can provide a better risk prediction compared to samples taken at a single time-point.

ELIGIBILITY:
Inclusion Criteria:

* Congenital Heart Disease Diagnosis
* Currently Pregnant

Exclusion Criteria:

* Unable to consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults (18+) who are currently pregnant
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Number of Subjects with cardiovascular adverse events | Baseline
  A cardiovascular adverse event is defined as Documented atrial/ventricular arrhythmias, need for cardioversion, arrhythmia-related procedures (catheter ablation, implantation of pacemaker/defibrillator, anti-arrhythmia surgery), and heart failure hospitalization.

SECONDARY OUTCOMES:
Number of Subject Deaths | Baseline
  Death will be determined as death due to end-stage heart failure, sudden cardiac death, thromboembolic death, and noncardiac death

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Egbe, MBBS, MPH, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No